CLINICAL TRIAL: NCT01167179
Title: Nurse-led Follow-up Care for Head and Neck Cancer Patients: a Quasi-experimental Study
Brief Title: Nurse-led Follow-up Care for Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Jacqueline de Leeuw, MSc, Radboud University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JDL-001-TVA
Record Dates: First submitted 2010-07-19; First posted 2010-07-22 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; nurse-led care; follow-up care; professional-patient relations; psychosocial adjustment; quasi-experimental; prospective; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- comparison group (No Intervention): Usual care Participants in the comparison group receive the usual care which consists of a 5 year medical routine control schedule based on the national guidelines, and - if appropriate - involvement of the dietician and the speech language therapist.During years one to five the routine control appointments are planned at a minimum of every 2, 3, 4, 6 and 12 months respectively. Most patients who undergo a total laryngectomy have additional contact with an oncology nurse during their 6-8 weekly medical control visits at the outpatient clinic for approximately the first year of follow-up. All other head and neck cancer patients have no structured follow-up contact with an oncology nurse.
- nurse-led consultation (Experimental): Interventional care Year 1 follow-up: 2-monthly medical control visit + 30 minute nursing consultation, to a minimum of 6 in year 1. No restrictions with regard to cancer stage, site or treatment modality.
  Intervention consist of standardised nursing consultations comprising a thorough needs assessment, supportive counseling, adequate referral to other care providers if necessary and improvement of the continuity of follow-up care. Goals: helping patients (and their partners) cope with the physical and psychosocial consequences of treatment and help them to gradually adjust to 'the life after', and into survivorship.
  Interventions: Behavioral: nurse-led consultation

INTERVENTIONS:
Behavioral: nurse-led consultation — Content of the intervention The intervention consists of structured and standardised nursing follow up consultations comprising a thorough needs assessment, supportive counseling, adequate referral to other care providers if necessary and improvement of the continuity of follow-up care. The goals of nursing follow-up care are summarised as helping patients (and often their partners too) to cope with the physical and psychosocial consequences of treatment and help them to gradually adjust to 'the life after', and into survivorship.
  Other Names: nurse-led follow-up care
  Arms: nurse-led consultation

SUMMARY:
The purpose of this study is to conduct an early evaluation of a nurse-led follow up intervention added to the usual medically oriented follow up care. Besides evaluating the feasibility and acceptability to patients, the effect on psychosocial adjustment and quality of life of patients is determined.

DETAILED DESCRIPTION:
Background: After treatment for cancer, follow-up surveillance is regarded important. In head and neck cancer patients however, increasing research evidence shows that at least the goal of detecting recurrence of cancer during routine control visits in an asymptomatic stage is not achieved. Other goals of follow-up such as management of treatment complications and helping patients and families cope and adjust remain important and ask for an accurate, effective but tailored and sensitive approach. Increasingly, nurses are mentioned as care providers best suited to perform this task.

Aim: The purpose of this study is to conduct an early evaluation of a nurse-led follow up intervention added to the usual medically oriented follow up care. Besides evaluating the feasibility and acceptability to patients, the effect on psychosocial adjustment and quality of life of patients is determined.

Methods and design: A quasi-experimental prospective design is used. Two groups of patients are enrolled consecutively (n=160) and patient data are collected at baseline (T0), at 6(T1) and at 12(T2) months respectively. The duration of the intervention is defined to the first year of follow up. Participating nurses are trained prior to the recruitment of the intervention group and receive supervision and individual coaching during the entire duration of the intervention phase.

Outcome measures: Primary outcome, psychosocial adjustment to illness. Secondary outcomes, health related quality of life, psychosocial problems, and usage of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a primary head and neck tumour
* Absence of other cancers diagnosed
* Treatment with curative intent, all treatment modalities
* Treatment and 12 month follow-up planned in Radboud University Nijmegen Medical Centre
* Able to speak, write and understand Dutch
* Cognitively able to give informed consent

Exclusion Criteria:

* Actual psychiatric disease
* Actual alcohol addiction
* Known life expectancy of < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T van Achterberg, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Leeuw J, Prins JB, Teerenstra S, Merkx MA, Marres HA, van Achterberg T. Nurse-led follow-up care for head and neck cancer patients: a quasi-experimental prospective trial. Support Care Cancer. 2013 Feb;21(2):537-47. doi: 10.1007/s00520-012-1553-1. Epub 2012 Aug 4. PMID 22864472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2007 to February 2010. Setting: outpatient oncology clinic
Pre-assignment Details: The eligibility criteria for the study were as follows: informed of a HNC diagnosis (but no other cancer); to be treated with curative intent; to be able to speak, write and understand Dutch; and be cognitively able to provide informed consent. Exclusion criteria included overt psychopathology, alcohol addiction, life expectancy of less than 6 mo.
Groups:
- Usual Care: The participants in the usual care group received care that consisted of a 5-year routine control schedule with six bimonthly 10-minute visits to a head and neck surgeon in the first year posttreatment in accordance with national guidelines.19 Nursing follow-up care consisted of ad hoc problem-based contacts except for patients who underwent a laryngectomy, who received standard nursing consultations during the first 6 months posttreatment in parallel with the medical control visits. Patients who were treated with surgery alone all had one standard wound control visit with a nurse; patients who were treated with radiotherapy had one to six ad hoc nursing contacts during the first 6 months posttreatment. For the duration of the study, there were no changes in usual care.
- Intervention: The intervention consisted of six 30-minute nursing follow-up consultations in the first year posttreatment. A standardized protocol was used for this purpose. Nursing consultations were conducted in parallel with and preceding the medical routine control visits and included a needs assessment based upon the biopsychosocial model.The aim of consultation was to give advice and support to patients (and their partners) addressing the physical and psychosocial consequences of treatment. To increase patient focus and active participation during consultations, patients completed a 13-item checklist prior to each consultation. Every 3 months, patients were screened for psychosocial problem areas using a specific questionnaire.
  During the consultations, the nurses also performed simple medical checks including inspection of the tracheal stoma, cannula and speech valve (if applicable), and oral cavity, and palpation of the neck and lymph nodes.
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 80 | 80
Completed | 65 | 59
Not Completed | 15 | 21
Not completed — disease recurrence | 4 | 4
Not completed — Death | 4 | 10
Not completed — Withdrawal by Subject | 1 | 2
Not completed — diverse | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: The participants in the comparison group received usual care that consisted of a 5-year routine control schedule with six bimonthly 10-minute visits to a head and neck surgeon in the first year posttreatment in accordance with national guidelines.19 Nursing follow-up care consisted of ad hoc problem-based contacts except for patients who underwent a laryngectomy, who received standard nursing consultations during the first 6 months posttreatment in parallel with the medical control visits. Patients who were treated with surgery alone all had one standard wound control visit with a nurse; patients who were treated with radiotherapy had one to six ad hoc nursing contacts during the first 6 months posttreatment. For the duration of the study, there were no changes in conventional care.
- Intervention: The intervention consisted of six 30-minute nursing follow-up consultations in the first year posttreatment. A standardized protocol was used for this purpose. Nursing consultations were conducted in parallel with and preceding the medical routine control visits and included a needs assessment based upon the biopsychosocial model. The aim of consultation was to give advice and support to patients (and their partners) addressing the physical and psychosocial consequences of treatment. To increase patient focus and active participation during consultations, patients completed a 13-item checklist prior to each consultation.Every 3 months, patients were screened for psychosocial problem areas using a specific questionnaire.During the consultations, the nurses also performed simple medical checks including inspection of the tracheal stoma, cannula and speech valve (if applicable), and oral cavity, and palpation of the neck and lymph nodes.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 69 | 137
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (13.0) | 59.2 (12.3) | 58.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 60 | 54 | 114
Region of Enrollment [Number; unit: participants]
  Netherlands | 80 | 80 | 160
Psychosocial adjustment [Mean (Standard Deviation); unit: units on a scale] — Psychosocial Adjustment to Illness Scale - Self Report (PAIS-SR), a 46-item self-report measure that assesses changes in seven domains. The Dutch validated questionnaire was used.HRQOL was measured with the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire with additional Head & Neck Module (EORTC QLQ-C30 and QLQ-H&N35).
  units on a scale | 46 (12) | 50 (11) | 49 (12)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Quality of Life(QoL)was measured with the EORTC QLQ-C30 and QLQ-H&N35.The EORTC QLQ-C30 contains five functioning scales, a global health status/QoL scale, and nine symptom scales. The QLQ-H&N35 contains 18 disease-specific symptom scales. All scores in both the EORTC QLQ-C30 and QLQ-H&N35 were transformed to a 0-100 scale following instructions in the scoring manual, with higher scores representing better quality of life and less disease-specific symptoms.
  units on a scale | 76 (17) | 64 (23) | 72 (19)

OUTCOME MEASURES:

1. Secondary Outcome: Quality of Life
Description: Quality of Life(QoL)was measured with the EORTC QLQ-C30 and QLQ-H&N35.The EORTC QLQ-C30 contains five functioning scales, a global health status/QoL scale, and nine symptom scales. The QLQ-H&N35 contains 18 disease-specific symptom scales. All scores in both the EORTC QLQ-C30 and QLQ-H&N35 were transformed to a 0-100 scale following instructions in the scoring manual, with higher scores representing better quality of life and less disease-specific symptoms.
Time Frame: baseline, 6 mo, 12 mo
Population: ITT analyses. Linear mixed model for repeated measurements.Intervention an time (as well as their interaction), and adjustment factors tumor location, size of the tumor,treatment modality, living without a partner, and education (high vs. other) were included in the model as fixed effects. An unstructured covariance matrix was fitted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 80 | 80
units on a scale
  baseline | 76 (17) | 64 (23)
  6 mo | 80 (18) | 77 (16)
  12 mo | 80 (17) | 81 (18)

2. Primary Outcome: Psychosocial Adjustment to Illness-Scale
Description: The adaptive psychosocial response of an individual to a significant life change was assessed using the Psychosocial Adjustment to Illness Scale -Self Report (PAIS-SR), a 46-item self-report measure that assesses changes in seven domains. A mean PAIS-SR T-score of 50 is the average score for each domain, meaning that patients with this score adjusted neither better nor worse than a mixed cancer reference group, whereas a score lower than 50 indicates better adjustment. The total scale range for the T score is 21-80. The PAIS-SR is well validated and has been used in previous studies of HNC patients.Here, we used the validated Dutch translation.
Time Frame: baseline, 6 mo, 12mo
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 80 | 80
units on a scale
  baseline | 46 (12) [43 to 60] | 50 (11)
  6 mo | 44 (12) | 44 (13)
  12 mo | 42 (12) | 43 (13)

ADVERSE EVENTS:
Arm/Group | Usual Care | Intervention
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

LIMITATIONS AND CAVEATS:
A historical control group being the comparison group was the 'usual care' group that included participants who were enrolled during the study and received usual care, as described.

Lack of randomization may have been a confounding factor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes